CLINICAL TRIAL: NCT03608501
Title: An Open-Label, Single-Arm Phase II Study of Ixazomib, Thalidomide and Dexamethasone in Newly Diagnosed and Treatment-Naive Multiple Myeloma Patients Non-Eligible for Autologous Stem-Cell Transplantation
Brief Title: A Study of Ixazomib, Thalidomide and Dexamethasone in Newly Diagnosed and Treatment-naive Multiple Myeloma (MM) Participants Non-eligible for Autologous Stem-cell Transplantation
Acronym: IDEALL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision (no safety or efficacy concerns)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16041; U1111-1214-1078 (Other: WHO)
Record Dates: First submitted 2018-07-11; First posted 2018-08-01 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Multiple Myeloma
Keywords: Drug therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ixazomib 4 mg + Thalidomide 100 mg + Dexamethasone 40 mg (Experimental): Ixazomib 4 milligram (mg), capsule, orally, once on Days 1, 8 and 15 along with thalidomide 100 mg, tablet, orally, once daily and dexamethasone 40 mg, tablet, orally, once on Days 1, 8, 15 and 22 in a 28-day treatment cycle for up to 9 cycles or until withdrawal from the study in the treatment phase. Participants who complete treatment phase will be eligible to continue on to the maintenance phase of the study to receive ixazomib 4 mg, capsules, orally, once on Days 1, 8 and 15 of a 28-day treatment cycle for up to 24 months or until withdrawal from the study.
  Interventions: Drug: Ixazomib; Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules.
  Other Names: Ixazomib citrate
Drug: Thalidomide — Thalidomide capsules.
Drug: Dexamethasone — Dexamethasone tablets.

SUMMARY:
The primary purpose of this study is to determine the overall response rate (ORR) during induction therapy with the combination of ixazomib, thalidomide and low-dose dexamethasone in specific time points.

DETAILED DESCRIPTION:
The drugs being tested in this study are a combination therapy of ixazomib, thalidomide and low-dose dexamethasone. This combination therapy is being tested to treat people who are newly diagnosed with multiple myeloma and non-eligible to autologous stem cell transplantation (ASCT). This study will assess the ORR during induction therapy in specific timepoints.

The study will enroll approximately 40 participants. All participants will receive:

Ixazomib citrate 4 mg + Thalidomide 100 mg and Dexamethasone 40 mg.

All participants will be asked to take their study medication at approximately the same time each day.

This multi-center trial will be conducted in Brazil. The overall time to participate in this study is approximately 5 years. Participants will make multiple visits to the clinic, and will be contacted by telephone or will make a final visit 30 days after receiving their last dose of drug or resolution of serious adverse event (SAE), whichever occurs later for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Clonal bone marrow plasma cells >=10% or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following myeloma defining events:

   * Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically:

     * Hypercalcaemia: serum calcium greater than (>) 1 mg/dL higher than the upper limit of normal (ULN) or >11 mg/dL;
     * Renal insufficiency: creatinine clearance <40 milliliter (mL) per minute (as per validated equations) or serum creatinine >2 mg/dL;
     * Anemia: haemoglobin value of >20 gram per liter (g/L) below the lower limit of normal, or a haemoglobin value <100 g/L;
     * Bone lesions: one or more osteolytic lesions on skeletal radiography, computed tomography (CT), or positron emission tomography (PET)-CT.
   * Any one or more of the following biomarkers of malignancy:

     * Clonal bone marrow plasma cell percentage >=60%.
     * Involved: uninvolved serum free light chain ratio >=100.
     * Greater than (>) 1 focal lesions on magnetic resonance imaging (MRI) studies. Note: clonality should be established by showing kappa to lambda ratio (κ/λ)-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate and core biopsy, the highest value should be used.
2. Ineligibility to autologous transplantation, as per investigator's discretion, regardless of age (the reason for such ineligibility should be recorded on the electronic case report form [eCRF]).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Ability to take concurrent aspirin daily (or enoxaparin subcutaneously daily), per published standard or institutional standard of care, as prophylactic anticoagulation.
5. Note: For participants with prior history of deep vein thrombosis (DVT), low molecular weight heparin (LMWH) is mandatory.
6. Left ventricular ejection fraction (LVEF) >=50%.
7. Clinical laboratory values as specified below within 7 days before the first dose of study drug:

   * Absolute neutrophil count (ANC) >=1,500 per cubic millimeter (/mm^3), unless related to bone marrow infiltration by malignant plasma cells.
   * Hemoglobin >=8.0 g/dL
   * Platelet count >=75,000/mm^3, unless related to bone marrow infiltration by malignant plasma cells (platelet transfusions to help participants meet eligibility criteria are not allowed).
   * Aspartate aminotransferase (AST) and alanine aminotransferase (AST) less than or equal to (<=) 1.5 times the institutional ULN.
   * Bilirubin <=1.5 mg/dL (or <=2.5 mg/dL in case of Gilbert-Meulengracht syndrome).
   * Glomerular filtration rate >=30 milliliter per minute per (mL/min/) 1.73 square meter (m^2) according to the Modification of Diet in Renal Disease (MDRD) study abbreviated formula. If not on target, this evaluation may be repeated once after at least 24 hours.
   * Prothrombin time (PT) or activated partial thromboplastin time (aPTT) within normal limits.

Exclusion Criteria:

1. Presence of non-secretory or oligo-secretory myeloma, smoldering MM, monoclonal gammopathy of undetermined significance, plasma-cell leukemia, Waldenstrom's macroglobulinemia, primary amyloidosis, or polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes (POEMS) syndrome.
2. Central nervous system involvement by MM.
3. Prior radiation therapy involving an estimated >=25% of the hematopoietically active bone marrow. Radiotherapy should not be given within 14 days before enrollment. In case of palliative radiotherapy for pain control and if the involved field is small, 7 days will be considered a sufficient interval between the radiation treatment and administration of the study drugs.
4. Treatment with any investigational products within 1 (one) year before the first dose of the study drug regimen.
5. Presence of peripheral neuropathy of grade 1 with pain or grade 2 or higher.
6. Previous or concurrent history of malignancies other than MM except for curatively treated cervical carcinoma in situ, non-melanoma skin cancer, superficial bladder cancer (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria]), or localized prostate cancer.
7. With evidence or history of bleeding diathesis. Any hemorrhage or bleeding event >=common terminology criteria for adverse events (CTCAE) Grade 3 within 4 weeks of start of study medication.
8. Major surgery within 14 days before randomization.
9. Non-healing wound or ulcer.
10. Seizure disorder requiring medication.
11. Systemic treatment with strong cytochrome P-450 3A (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort from Day-14 of cycle 1 until the safety follow-up.
12. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
ORR During Induction | Upon ORR assessment during specific timepoints for all participants completing or withdrawn prematurely from the induction phase (Baseline up to approximately 9 month [Cycle 9])
  ORR is the percentage of participants with presence of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR). ORR assessment will be based on International Myeloma Working Group (IMWG) response criteria.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Upon study termination (Baseline up to first documentation of disease progression [PD] or death from any cause [approximately 2 years])
  PFS is the time elapsed between treatment initiation and first PD documentation or death from any cause, where PD is assessed by IMWG response criteria.
ORR During Maintenance | Upon ORR assessment during specific time points for all participants completing or withdrawn prematurely from maintenance phase (Baseline up to approximately 2 years)
  ORR is the percentage of participants with presence of sCR, CR, VGPR or PR. ORR assessment will be based on IMWG response criteria.
Overall Survival (OS) | Upon study termination (Baseline up to approximately 5 years)
  OS is defined as the time elapsed between treatment initiation and death from any cause.
Time to Response During Induction | End of induction phase (Baseline up to approximately 9 months [Cycle 9])
  Time to response is the time elapsed between treatment initiation and the first documentation of sCR, VGPR or PR according to the IMWG response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (6):
- Brazil (6):
  - CEHON Centro de Hematologia e Oncologia da Bahia, Salvador, Estado de Bahia
  - Instituto COI de Educacao e Pesquisa, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Estadual de Campinas UNICAMP - HEMOCENTRO, Campinas, São Paulo
  - Clinica Medica Sao Germano S/S Ltda., São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.